CLINICAL TRIAL: NCT05573074
Title: Transcranial Near Infrared Radiation and Cerebral Blood Flow in Depression - R33
Acronym: TRIADE-R33
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 22-01065
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: MDD, transcranial Photobiomodulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tPBM Group (Experimental): Visit 1: t-PBM at irradiance dose of 291.7 mW/cm2 (333s) Visit 2 - 18: randomized to receive active t-PBM of 291.7 mW/cm2 (333s) Visit 19: t-PBM at irradiance dose of 291.7 mW/cm2 (333s)
  Interventions: Device: Transcranial Photobiomodulator; Device: Sham
- Sham Group (Active Comparator): Visit 1: t-PBM at irradiance does of 291.7 mW/cm2 (333s) Visit 2 - 18: randomized to receive Sham of 0 mW/cm2 (333s) Visit 19: t-PBM at irradiance dose of 291.7 mW/cm2 (333s)
  Interventions: Device: Transcranial Photobiomodulator; Device: Sham

INTERVENTIONS:
Device: Transcranial Photobiomodulator — Transcranial photobiomodulator delivers Near-Infrared Radiation (NIR) continuous middle irradiance (291.7 mW/cm2) to patients' foreheads.
  Other Names: LightForce EXPi tPBM-2.0
Device: Sham — Transcranial Photobiomodulator delivers sham irradiance odes of 0 mW/cm2

SUMMARY:
The purpose of this research study is to determine if application of near infrared energy to the forehead can change blood flow in the brains of people with depression. Near infrared energy is like light but is not visible to the human eye.

DETAILED DESCRIPTION:
In this multi-center study, approximately 60 subjects with Major Depressive Disorder (MDD) will undergo Magnetic Resonance Imaging (MRI) scanning during transcranial Photobiomodulation (tPBM) before and after a randomized, double-blinded, controlled 16 session course of treatment with tPBM or sham.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to give written informed consent and follow study procedures
* Participants must be 18-65 years of age
* Participants must have major depressive disorder; all the following conditions need to be met to ensure presence of significant depression symptoms:

  1. Meeting diagnostic criteria for Major Depressive Disorder (MDD) in the past two weeks, at the DSM-5 Mini-International Neuropsychiatric Interview (MINI)
  2. Inventory for Depressive Symptomatology Clinician-rated (IDS-C) total score ≥23 at screening
  3. Depression symptoms are the primary target of treatment or treatment-seeking.
* Women of child-bearing potential must agree to use adequate contraception
* Participants taking medications or psychotherapy approved for the treatment of major depressive disorder will need to be stable for at least 8 weeks prior to screen.

Exclusion Criteria:

* Unwilling or unable to comply with study requirements
* Patients judged to be at serious and imminent suicidal (C-SSRS≥4) or homicide risk, or currently in crisis such that inpatient hospitalization or other crisis management should take priority.
* History of any or psychotic or bipolar disorder
* Met diagnostic criteria for an alcohol or substance use disorder, post-traumatic stress disorder, obsessive-compulsive disorder, anorexia nervosa, or bulimia nervosa within the preceding 6 months
* History of dementia, traumatic brain injury (TBI), or neurological disorders affecting the brain, including any history of stroke or seizure disorders requiring treatment in the last 5 years
* Cognitive impairment significant as determined by the Montreal Cognitive Assessment (MOCA) <22 or MOCA-Blind <19.
* History of antisocial personality disorder, or any clinically significant personality trait that would, in the investigator's judgment, preclude safe study participation or impair ability to remain adherent with the treatment protocol
* History of significant treatment non-adherence or situations where the subjects are unlikely to adhere to treatment, in the opinion of the investigator.
* Pregnant (as confirmed by pregnancy test at screen) or nursing
* Currently undergoing device-based treatment for depression or taking medications for depression other than SSRIs, SNRIs, or Wellbutrin (bupropion).
* Treatment resistance with failure to respond to more than two adequate treatments with FDA-approved antidepressant medications during current episode of major depressive disorder.
* History of ECT in the last 12 months; lifetime history of VNS; lifetime treatment resistance to any FDA-approved device-based treatment for major depressive disorder (such as ECT, TMS, VNS); device-based interventions for depression will need to be discontinued at least 8 weeks prior to screen.
* Serious, unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, hematologic disease; defined as any medical illness which is not well-controlled with standard-of-care v Clinically significant abnormal findings of laboratory parameters including urine toxicology screen for drugs of abuse or at physical examination.
* Clinical or laboratory evidence of uncontrolled hypothyroidism; if maintained on thyroid medication must be euthyroid for at least 1 month before screening.
* Past intolerance or hypersensitivity to tPBM.
* Significant skin conditions (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that are found in the area of the procedure sites.
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.
* Any type of implants in the head, whose functioning might be affected by tPBM (e.g., stent, clipped aneurysm, embolized AVM, implantable shunt - Hakim valve).
* Failure to meet standard MRI safety requirements (e.g., claustrophobia, non-removable piercings, implanted medical devices, other non-removable metals) as determined by the MRI Safety Checklist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent change of cerebral blood flow (CBF) | Baseline, Visit 18 (Week 10)
  Cerebral blood flow (CBF) is measured as Blood oxygen Level Dependent (BOLD) signal on functional magnetic resonance imaging (fMRI). BOLD signal reflect changes in regional cerebral blood flow that delineates regional activity, A positive BOLD signal marks an increase in regional blood flow while a negative BOLD signal marks a decrease in regional blood flow. A positive percent change indicates that blood flow increased in the region of interest between scans, a negative percent change indicates blood flow decreased between scans.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 17 (Week 9, endpoint)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.

SECONDARY OUTCOMES:
Percent change of cerebral blood flow (CBF) at endpoint in relation to treatment outcome | Baseline, Visit 18 (Week 10)]
  Cerebral blood flow (CBF) is measured as Blood oxygen Level Dependent (BOLD) signal on functional magnetic resonance imaging (fMRI). BOLD signal reflect changes in regional cerebral blood flow that delineates regional activity, A positive BOLD signal marks an increase in regional blood flow while a negative BOLD signal marks a decrease in regional blood flow. A positive percent change indicates that blood flow increased in the region of interest between scans, a negative percent change indicates blood flow decreased between scans. Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression. MADRS change score from baseline to endpoint
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 3 (Week 2)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 5 (Week 3)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 7 (Week 4)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 9 (Week 5)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 11 (Week 6)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 13 (Week 7)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, Visit 15 (Week 8)
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Harvard Medical School, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request, Requests should be directed to dan.iosifescu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement